CLINICAL TRIAL: NCT04952948
Title: Effect of Short Period of Detraining of the Pilates Method on Functional Capacity and Blood Pressure of Elderly Women With Type 2 Diabetes
Brief Title: Pilates Method on Functional Capacity and Blood Pressure of Elderly Women With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do vale do São Francisco (Other)
Responsible Party: Principal Investigator, Sérgio Rodrigues Moreira, Professor (PhD), Universidade Federal do vale do São Francisco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4
Record Dates: First submitted 2021-06-11; First posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Type-2 Diabetes; Physical Disability; Blood Pressure
Keywords: Resistance exercise; Functionality; Interruption; Diabetes; Cardiovascular
MeSH Terms: conditions — Diabetes Mellitus | interventions — Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PILATES Method Training Group (Experimental): The PILATES program at moderate intensity lasted 12 weeks, at a frequency of 3 times a week, and with duration of 60 minutes for each exercise session.
  Interventions: Other: PILATES Training
- CONTROL Group (Sham Comparator): While the PILATES Group participated in the intervention with physical exercises, the CONTROL group only participated in the functional capacity and blood pressure assessments. However, at the end of the intervention in the PILATES Group, the CONTROL Group was invited to participate in a similar training program.
  Interventions: Other: PILATES Training

INTERVENTIONS:
Other: PILATES Training — During the PILATES sessions, the practitioner received orientations to to perform slow movements, aware, and combined with the respiratory cycle. The exercises program was performed on a soft ground covered with tatamis. During the program, a set of swiss balls of 45, 55, and 65 cm in size and elastic bands of very moderate resistance were used. Each exercise session was divided into 3 stages, namely (a) global initial static and dynamic stretching (10 minutes); (b) general conditioning (45 minutes) and; (c) relaxation (5 minutes). The amount of series and repetitions per set in exercises, in addition to the intensity required in each session in PILATES is presented in Table 2 of Melo et al. (2020) - Vide reference.

SUMMARY:
Type 2 diabetes mellitus (T2D) is a chronic inflammatory disease that is associated with loss of functional capacity and increased blood pressure. Coupled with this, there is an increased risk of falls and fractures in patients with T2D. On the other hand, conventional training programs for resistance, aerobic or combined exercises are strongly recommended for people with T2D, as they promote a reduction in the glycemic rate and blood pressure, and an improvement in functional capacity. However, little is known about unconventional training programs such as PILATES (dynamic and isometric muscle actions) on functional capacity and cardiovascular adaptations in T2D.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2D) is a chronic inflammatory disease whose main mechanism of installation is insulin resistance and is associated with loss of functional capacity with consequent fragility and increased blood pressure. Currently, women have the highest prevalence of T2D in Brazil. Previous studies have shown that women are more affected by cases of hospitalization and that they have a higher risk of mortality due to illness. Muscle function and strength in patients with T2D show a reduction compared to healthy and normoglycemic subjects, especially in menopausal women, when estrogen declines with a consequent increase in body fat and decreased muscle quality. Coupled with this, there is a reduction in muscle mass and an increased risk of falls and fractures in patients with T2D. Its association with other factors such as physical inactivity, involuntary weight loss, less muscle strength and slower gait can lead to frailty and limit the performance of basic daily activities. On the other hand, conventional training programs for resistance, aerobic or combined exercises are strongly recommended for people with T2D, as they promote a reduction in the glycemic rate and blood pressure, and an improvement in functional capacity. Unconventional training programs such as PILATES (dynamic and isometric muscle actions) ensure the control of forces that act on the musculoskeletal system, promoting an important improvement in functional capacity and possible cardiovascular adaptations. Additionally, elderly people have pronounced losses of neuromuscular adaptations even in a short period of detraining, compromising gains related to functional capacity and this loss can be even more pronounced in patients with T2D. Therefore, it is also necessary for training professionals to understand the effects of the short detraining period after unconventional exercise programs like PILATES on the functional capacity of elderly women with T2D as well as to understand the effects of the PILATES training on blood pressure or cardiovascular adaptations.

ELIGIBILITY:
Inclusion Criteria:

* Present a diagnosis of type-2 diabetes;
* Do not have severe or decompensated heart disease;
* Do not have coronary artery disease;
* Do not have peripheral neuropathy and ulcers in the extremities;
* Do not have severe skin lesions;
* Do not have proliferative retinopathy;
* Do not have insulin therapy;
* Do not have any health condition that would hinder participation in the exercise sessions.

Exclusion Criteria:

* Present some unexpected abnormality in health conditions during the research;
* Do not participate in more than 80% of the training sessions in the PILATES group.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-08-23 (Actual); Primary Completion 2016-11-28 (Actual); Study Completion 2016-12-19 (Actual)

PRIMARY OUTCOMES:
Change in functional capacity in type-2 diabetes | Pre-intervention (week zero) versus 4 weeks of intervention in PILATES Group and CONTROL group
  Measurements of functional capacity (time in seconds of execution of the functional tests) in the PILATES and CONTROL groups to be analyzed in the pre-intervention and post-intervention moments.
Change in functional capacity in type-2 diabetes | Pre-intervention (week zero) versus 8 weeks of intervention in PILATES Group and CONTROL group
  Measurements of functional capacity (time in seconds of execution of the functional tests) in the PILATES and CONTROL groups to be analyzed in the pre-intervention and post-intervention moments.
Change in functional capacity in type-2 diabetes | Pre-intervention (week zero) versus 12 weeks post-intervention in PILATES Group and CONTROL group
  Measurements of functional capacity (time in seconds of execution of the functional tests) in the PILATES and CONTROL groups to be analyzed in the pre-intervention and post-intervention moments.
Change in functional capacity in type-2 diabetes | Pre-intervention (week zero) versus 4 weeks of detraining post-intervention in PILATES Group and CONTROL group
  Measurements of functional capacity (time in seconds of execution of the functional tests) in the PILATES and CONTROL groups to be analyzed in the pre-intervention and detraining moments.
Change in functional capacity in type-2 diabetes | Pos-intervention (12 weeks) versus 4 weeks of detraining (4W_DT) in PILATES Group and CONTROL group
  Measurements of functional capacity (time in seconds of execution of the functional tests) in the PILATES and CONTROL groups to be analyzed in the post-intervention and detraining moments.
Change in blood pressure in type-2 diabetes | Pre-intervention (week zero) versus 4 weeks of intervention in PILATES Group and CONTROL group
  Measurements of systolic blood pressure and diastolic blood pressure (mmHg) in the PILATES and CONTROL groups to be analyzed in the pre-intervention and post-intervention moments.
Change in lood pressure in type-2 diabetes | Pre-intervention (week zero) versus 8 weeks of intervention in PILATES Group and CONTROL group
  Measurements of systolic blood pressure and diastolic blood pressure (mmHg) in the PILATES and CONTROL groups to be analyzed in the pre-intervention and post-intervention moments.
Change in blood pressure in type-2 diabetes | Pre-intervention (week zero) versus 12 weeks post-intervention in PILATES Group and CONTROL group
  Measurements of systolic blood pressure and diastolic blood pressure (mmHg) in the PILATES and CONTROL groups to be analyzed in the pre-intervention and post-intervention moments.

CONTACTS AND LOCATIONS:
Overall Officials: Ilka Yolane TP Andrade, Ms, Study Chair — Federal University of Vale do São Francisco - UNIVASF

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Melo KCB, Araujo FS, Cordeiro Junior CCM, de Andrade KTP, Moreira SR. Pilates Method Training: Functional and Blood Glucose Responses of Older Women With Type 2 Diabetes. J Strength Cond Res. 2020 Apr;34(4):1001-1007. doi: 10.1519/JSC.0000000000002704. PMID 29985228